CLINICAL TRIAL: NCT04754919
Title: Study Into the Use of a Diabetes Specialist Transition Nurse in the Care of Young People With Type 1 Diabetes Undergoing Transition From the Paediatric to the Adult Services, at the Northampton General Hospital
Brief Title: The Diabetes Transition Study for Young People Aged Between 16-20 Years of Age.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northampton General Hospital NHS Trust (Other)
Responsible Party: Principal Investigator, Dr Anne Smith, Consultant Paediatrician, Northampton General Hospital NHS Trust
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 10087
Record Dates: First submitted 2019-08-22; First posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Next 50 eligible young people entering transition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transition intervention group (Active Comparator): Intervention group -will be working with the specialist diabetes transition nurse. The nurse will follow a specific protocol involving visits, clinic support, community support and appointment rearranging. She will also maintain communication with the Hospital based adult and paediatric diabetes teams and the participants General Practitioner and relevant community health care professionals.
  Interventions: Other: Transition intervention group
- Post Transition group (Placebo Comparator): The previous fifty eligible young people who have transitioned to adult service, will be compared with the active comparator group.
  Interventions: Other: Post transition group

INTERVENTIONS:
Other: Transition intervention group — Support and on-going treatment intervention; monitoring the uptake of routine annual diabetes tests and encouraging to access where default observed General specialist diabetes support and provision of education and referral to other specialist healthcare agencies as individual requires
  Arms: Transition intervention group
Other: Post transition group — The previous fifty eligible young people who have transitioned to adult service, will be compared with the active comparator group.
  Arms: Post Transition group

SUMMARY:
Study into the use of a diabetes specialist transition nurse in the care of young people aged 16-20 years, with type 1 diabetes; undergoing transition from the paediatric to the adult diabetes services at the Northampton General Hospital

DETAILED DESCRIPTION:
Does the use of a structured diabetes transition program in the care of young people transitioning from the paediatric to the adult diabetes services at Northampton General Hospital improve the study group mean HbA1C, reduce the number of diabetes related hospital episodes and increase attendance at the adult diabetes clinic following transition to the adult service?

ELIGIBILITY:
Inclusion Criteria:

* established type 1 diabetes for minimum of 1 year
* attended the Northampton general Hospital, children's and young peoples diabetes service for at least 6 months prior to transition
* between the ages of 16 - 20 years
* ability to participate in all aspects of the trial
* written informed consent must be obtained

Exclusion Criteria:

* any condition which may interfere with the subjects ability to participate in the study including cystic-fibrosis related diabetes
* subjects who move away from the Northampton General Hospital clinic during the transition process
* those unable to give informed consent

Ages: 16 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
The rates of diabetes related hospital episodes, including Diabetic Ketoacidosis, between the 2 study groups before and after transition | 3 years
  Rates of admission

SECONDARY OUTCOMES:
The mean Hba1C between the 2 study groups before and after transition | 3 years
  Hba1C measurement
The frequency of testing according to National Institute for Health and Care Excellence between the 2 study groups | 3 years
  Annual diabetes routine checks
Emotional health of the 2 study groups | 3 years
  HADS Questionnaire
Emotional health of the 2 study groups | 3 years
  PAID Questionnaire
To compare the proportion of young people in the study groups who fail to attend at least one out-patient adult diabetes appointment during the first year after transition | 3 years
  Compare attendance rates

CONTACTS AND LOCATIONS:
Overall Officials: Anne L Smith, MBChB, Principal Investigator — Northampton General Hospital
Locations (1):
- Northampton general Hospital NHS Trust, Northampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data, with other researchers

REFERENCES:
- [Result] Crowley R, Wolfe I, Lock K, McKee M. Improving the transition between paediatric and adult healthcare: a systematic review. Arch Dis Child. 2011 Jun;96(6):548-53. doi: 10.1136/adc.2010.202473. Epub 2011 Mar 8. PMID 21388969
- [Result] Spaic T, Mahon JL, Hramiak I, Byers N, Evans K, Robinson T, Lawson ML, Malcolm J, Goldbloom EB, Clarson CL; JDRF Canadian Clinical Trial CCTN1102 Study Group. Multicentre randomized controlled trial of structured transition on diabetes care management compared to standard diabetes care in adolescents and young adults with type 1 diabetes (Transition Trial). BMC Pediatr. 2013 Oct 9;13:163. doi: 10.1186/1471-2431-13-163. PMID 24106787
- See also: National Institute for Health and Care Excellence guidance adults — http://www.nice.org.uk/guidance/ng17
- See also: National Institute for Health and Care Excellence guidance for children and young people — http://www.nice.org.uk/guidance/ng18
- See also: Problem Areas in Diabetes Questionaire — http://www.researchgate.net/publication/7588148